CLINICAL TRIAL: NCT02037711
Title: Intraperitoneal Instillation of Levobupivacaine in Laparoscopic Pediatric Procedures
Brief Title: Intraperitoneal Application of Levobupivacaine During Laparoscopic Surgery in Kids.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif Mohamed Abd el moneim Soaida, MD, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: SMS2013
Record Dates: First submitted 2013-12-23; First posted 2014-01-16 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Pain
Keywords: Laparoscopic; Levobupivacaine; Pediatric; Anesthesia; Instillation; surgeries
MeSH Terms: conditions — Pain | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chirocaine group (levobupivacaine ) (Active Comparator)
  Interventions: Drug: Levobupivacaine 0.5%
- Control group (Sham Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Levobupivacaine 0.5% — Group I (Chirocaine group) (n=20): Levobupivacaine 0.5% will be instilled during insufflations of CO2 at the beginning of surgery at a dose of 2mg/kg.
  Arms: Chirocaine group (levobupivacaine )
Drug: Normal saline — Group II (control group) (n=20): laparoscopy done with instillation of normal saline instead of levobupivacain
  Arms: Control group

SUMMARY:
Pain after laparoscopic surgery has been associated with surgical manipulations, including intraperitoneal insufflation of carbon dioxide (CO2), resulting in peritoneal stretching, diaphragmatic irritation, changes in intra-abdominal pH, and retention of the insufflated gas in the abdominal cavity after surgery. These effects may result in the irritation of peritoneal nerves causing visceral pain, as commonly reported after laparoscopic procedures in pediatrics.

The study hypothesis is that Intraperitoneal local anesthetic (levobupivacaine) instillation can provide pain relief after laparoscopic surgery, but local anesthetic distribution may not always be uniform throughout the peritoneal surface. Many methods were tried for intraperitoneal application of local anesthetics in laparoscopic surgery such as local anesthetic (LA) instillation and LA nebulization.

-But these methods are not widely used in pediatrics upon our knowledge

ELIGIBILITY:
Inclusion Criteria:

1. Patient undergoing laparoscopic surgeries
2. Pediatric weighing 4 kg or more
3. Patients with free medical history

Exclusion Criteria:

1. Parents refusal
2. Known allergy to levobupivacaine
3. Acute preoperative pain other than biliary colic
4. chronic pain treatment or antiepileptic therapy
5. Severe hepatic or renal impairment
6. Cognitive impairment or communication problems.

Max Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2013-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain scoring (CHEOPS) | up to six hours
  pain score will be assessed immediately postoperative, then after 1 hour, 2 hours, and 6 hours.

SECONDARY OUTCOMES:
changes in Haemodynamics including ( Heart Rate) | during the period of the operation (Preoperative, post-induction, after instillation of levobupivacaine or saline, postoperative for 6 hours at 0-1-2-6
  Represented as mean and standard deviation, hemodynamic variables will be measured during the the surgery starting preoperatively, following induction of anesthesia, during the procedure and postoperatively (6 hours postoperative)
changes in Haemodynamics including ( Non Invasive Blood Pressure) | during the period of the operation (Preoperative, post-induction, after instillation of levobupivacaine or saline, postoperative for 6 hours at 0-1-2- 6
  Represented as mean and standard deviation, hemodynamic variables will be measured during the the surgery starting preoperatively, following induction of anesthesia, during the procedure and postoperatively (6 hours postoperative)

OTHER OUTCOMES:
Indirect signs of local anaesthetic toxicity (intraoperative arrhythmias and delayed awakening) | From time of instillation of levobupivacaine till 6 hours postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Saad El Basha, M.D., Study Chair — Cairo University; Maha Gmail, M.D., Study Director — Cairo University; Sherif M Soaida, M.D., Study Director — Cairo University; hagar H Refaee, Principal Investigator — Cairo University
Locations (1):
- Faculty of medicine, Cairo University, Cairo, Egypt